CLINICAL TRIAL: NCT05991882
Title: Mobile Adaptive Intervention to Reduce Negative Consequences Associated With Simultaneous Alcohol and Marijuana Use in Young Adults in Primary Care
Brief Title: Mobile Intervention for Simultaneous Alcohol and Marijuana Use in Young Adults
Acronym: SAFERR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R34DA056759 (NIH); R34DA056759 (NIH)
Record Dates: First submitted 2023-05-01; First posted 2023-08-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Drinking; Cannabis Use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of eight conditions
Who Masked: Participant
Masking Description: Participants in the factorial trial will be informed generally of the assigned condition (i.e., introduction module + no daily messages or introduction module + daily messages), but not given detailed content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Condition 1: Craving daily+PBS daily (Experimental): EMA + Introduction Module + Craving reduction and protective behavioral strategy (PBS) messages, each delivered once daily
  Interventions: Behavioral: Condition 1: Craving daily+PBS daily
- Condition 2: Craving daily+PBS trigger (Experimental): EMA + Introduction Module + Craving reduction messages delivered once daily and PBS trigger messages
  Interventions: Behavioral: Condition 2: Craving daily+PBS trigger
- Condition 3: Craving trigger+PBS daily (Experimental): EMA + Introduction Module + Craving reduction trigger messages and PBS messages delivered once daily
  Interventions: Behavioral: Condition 3: Craving trigger+PBS daily
- Condition 4: Craving trigger+PBS trigger (Experimental): EMA + Introduction Module + Craving reduction trigger and PBS trigger messages
  Interventions: Behavioral: Condition 4: Craving trigger+PBS trigger
- Condition 5: PBS daily+ PBS trigger (Experimental): EMA + Introduction Module + PBS delivered once daily and PBS trigger messages
  Interventions: Behavioral: Condition 5: PBS daily+ PBS trigger
- Condition 6: Craving daily+Craving trigger (Experimental): EMA + Introduction Module + Craving reduction delivered once daily and craving reduction trigger messages
  Interventions: Behavioral: Condition 6: Craving daily+Craving trigger
- Condition 7: Craving daily+Craving trigger+PBS daily+PBS trigger (Experimental): EMA + Introduction Module + Craving reduction delivered once daily, craving reduction trigger messages, PBS delivered once daily, and PBS trigger messages
  Interventions: Behavioral: Condition 7: Craving daily+Craving trigger+PBS daily+PBS trigger
- Condition 8: No daily or trigger craving or PBS (Other): EMA + Introduction Module + no other messages
  Interventions: Behavioral: Condition 8: No daily or trigger craving or PBS

INTERVENTIONS:
Behavioral: Condition 1: Craving daily+PBS daily — Participants in this condition will complete ecological momentary assessment (EMA) for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will then receive craving reduction and protective behavioral strategy (PBS) messages, each delivered once daily, until the end of the six-week period.
  Arms: Condition 1: Craving daily+PBS daily
Behavioral: Condition 2: Craving daily+PBS trigger — Participants in this condition will complete EMA for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will then receive craving reduction messages delivered once daily and PBS trigger messages that will be based on responses to signal-contingent EMA questions.
  Arms: Condition 2: Craving daily+PBS trigger
Behavioral: Condition 3: Craving trigger+PBS daily — Participants in this condition will complete EMA for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will then receive craving reduction messages that will be delivered based on responses to signal-contingent EMA questions and PBS delivered once daily.
  Arms: Condition 3: Craving trigger+PBS daily
Behavioral: Condition 4: Craving trigger+PBS trigger — Participants in this condition will complete EMA for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will then receive craving reduction and PBS messages delivered based on responses to signal-contingent EMA questions.
  Arms: Condition 4: Craving trigger+PBS trigger
Behavioral: Condition 5: PBS daily+ PBS trigger — Participants in this condition will complete EMA for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will then receive PBS messages delivered once daily and PBS trigger messages that will be based on responses to signal-contingent EMA questions.
  Arms: Condition 5: PBS daily+ PBS trigger
Behavioral: Condition 6: Craving daily+Craving trigger — Participants in this condition will complete EMA for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will then receive craving reduction messages delivered once daily and craving reduction trigger messages that will be based on responses to signal-contingent EMA questions.
  Arms: Condition 6: Craving daily+Craving trigger
Behavioral: Condition 7: Craving daily+Craving trigger+PBS daily+PBS trigger — Participants in this condition will complete EMA for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will then receive craving reduction and PBS messages delivered once daily and non-repetitive craving reduction and PBS trigger messages that will be based on responses to signal-contingent EMA questions.
  Arms: Condition 7: Craving daily+Craving trigger+PBS daily+PBS trigger
Behavioral: Condition 8: No daily or trigger craving or PBS — Participants in this condition will complete EMA for six weeks. Following the initial two weeks of EMA, participants in this condition will complete an introduction module including psychoeducation, personalized feedback, and goal setting. Participants will not receive any further intervention strategies.
  Arms: Condition 8: No daily or trigger craving or PBS

SUMMARY:
The goal of this treatment development project is to develop an adaptive ecological momentary intervention (a-EMI) for young adults using marijuana and alcohol that is grounded in self-regulation and social cognitive theories. To determine the most efficacious intervention strategies, the investigators will test variations of intervention components to identify the best combination. The study will take place at the Center for Integrated Health Care Research at Kaiser Permanente Hawaii (KPHI), located in Honolulu (island of Oahu). Following pilot testing with 6 participants, the study team will assess the feasibility and efficacy of intervention components on two primary outcomes (negative consequences and protective behavioral strategies [PBS]) using a fractional factorial experimental design, with post-intervention assessment and one- and three-month follow-ups. 136 diverse young adults recruited from KPHI who report current simultaneous alcohol and marijuana (SAM) use will be randomly assigned to one of eight groups, representing experimental conditions that include or do not include intervention strategies focused on craving reduction and PBS. As a result of this process, individual and/or combined components that lead to improved outcomes will be retained in a subsequent randomized controlled trial, while ineffective components will be eliminated.

DETAILED DESCRIPTION:
Up to one-third of young adults report use of marijuana or alcohol in the past month, with sizable numbers reporting daily marijuana use and heavy episodic drinking. Simultaneous alcohol and marijuana (SAM) use, defined as use of both substances at the same time or within a few hours of each other with overlapping effects, is common among young adults. Recent research has shown that SAM use leads to greater negative consequences compared to use of either substance alone. No current intervention addresses SAM use specifically and few leverage new technological methods (e.g., smartphones) or strategies (e.g., protective behavioral strategies [PBS]) to engage young adults.

The goal of this Stage I treatment development project is to develop a fully mobile adaptive ecological momentary intervention (a-EMI) titled "Smartphone App For Effectively Reducing Risk (SAFERR)" that is grounded in self-regulation and social cognitive theories. To determine the most efficacious intervention strategies, the investigators will test variations of intervention components to identify the best combination. They will assess the feasibility and efficacy of intervention components on two outcomes (negative consequences and PBS) using a fractional factorial experimental design.

The study will take place at the Center for Integrated Health Care Research at Kaiser Permanente Hawaii (KPHI), located in Honolulu (island of Oahu). Following pilot testing, the SAFERR a-EMI will be administered to 6 eligible participants. Based on the feedback, the app will be revised and a trial of the SAFERR intervention will begin. 136 diverse young adults who report current SAM use will be recruited from primary care clinics at KPHI. Eligible individuals will complete a baseline assessment and then be randomly assigned (by sex) to one of eight conditions using stratified randomization. Each condition either includes or does not include four different intervention strategies focused on craving reduction and PBS. All participants will complete signal-contingent (random prompts three times per day) and event-related ecological momentary assessment (EMA) for 6 weeks using a smartphone application (app). EMA will continue during the 4-week intervention phase. At the beginning of the intervention, all participants will complete an introduction module via the study app that includes psychoeducation, personalized feedback, and goal setting. Participants will then begin the a-EMI via the study app, with components delivered based on their condition assignment.

Following completion of the intervention, participants will complete a post-intervention assessment and follow-up assessments at one- and three-months. The feasibility of the a-EMI and design will be examined by assessing: study attrition and response rates/time, module completion rates, acceptability (satisfaction, usability), perceived helpfulness, goal attainment, and implementation and intervention engagement. The efficacy of intervention components on negative consequences and PBS during EMA and at post-intervention and one-month and three-month follow-ups will be examined. In a future, larger study, the most useful components will be incorporated into a full intervention package and tested in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* resident of state of Hawai'i and island of O'ahu
* age 18-30 years
* has sought services at Kaiser Permanente Hawaii within the past year
* report marijuana use, heavy drinking, and simultaneous alcohol and marijuana use
* report confidence in ability to use protective behavioral strategies
* endorse at least 3 recent negative consequences from marijuana and/or alcohol
* own a smartphone

Exclusion Criteria:

• any substance use treatment within the past 3 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Negative consequences associated with alcohol, marijuana, and simultaneous alcohol and marijuana (SAM) use | Through study completion, an average of 5 months
  Changes in negative consequences will be assessed using a measure that assesses alcohol, marijuana, and SAM use negative consequences. Items are rated dichotomously (yes/no).
Protective behavioral strategies for alcohol | Through study completion, an average of 5 months
  Changes in protective behavioral strategies for alcohol will be assessed using the Protective Drinking Practices Scale (PDPS), which assesses use of protective behavioral strategies related to alcohol on a 1 (never) to 6 (always) scale.
Protective behavioral strategies for marijuana | Through study completion, an average of 5 months
  Changes in protective behavioral strategies for marijuana will be assessed using the Protective Behavioral Strategies for Marijuana (PBSM) Scale, which assesses use of protective behavioral strategies related to marijuana on a 1 (never) to 6 (always) scale.

SECONDARY OUTCOMES:
Feasibility - study attrition | Through study completion, an average of 5 months
  Number of completed study phases, including six weeks of ecological momentary assessment (EMA), the 4-week a-EMI period, post-intervention assessment, and one- and three-month follow-up assessments.
Feasibility - response rate | Week 7
  Number of completed prompts across 6-week EMA
Feasibility - module completion rate | Week 7
  Completion of introduction module focused on psychoeducation, personalized feedback, and goal setting
Feasibility - acceptability of the intervention | Week 7
  The revised Client Satisfaction Questionnaire (CSQ-8) will assess satisfaction with the intervention, perceptions of format and language of the a-EMI messages, and usability of the a-EMI (e.g., manner in which information was presented, language, question/intervention strategy comprehension, strategy delivery, timing, and study and a-EMI burden).
Feasibility - perceived helpfulness of intervention strategies | Week 7
  A Feedback Measure will assess perceptions of the helpfulness of particular intervention strategies, as well as other useful strategies that could be added.
Feasibility - intervention implementation | Week 7
  Intervention implementation will be examined through a short survey that will assess the ease of app use and accessibility, any challenges requesting strategies when needed, and any problems with the technology.
Feasibility - intervention engagement | Week 7
  Intervention engagement will be assessed by examining participant's use of intervention strategies.
Feasibility - goal attainment | Through study completion, an average of 5 months
  Participants will be asked to report whether they attained or made progress on goals identified in the a-EMI introduction module.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Phillips, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Hawaii, Center for Integrated Health Care Research, Honolulu, Hawaii, United States